CLINICAL TRIAL: NCT03043495
Title: The Optimal Dose Of Dexamethasone To Be Used As An Adjuvant To Low Volume Bupivacaine Ultrasound Guided Supraclavicular Brachial Plexus Block. A Randomized Controlled Double Blinded Dose Ranging Study
Brief Title: Dexamethasone Dose in Low Volume Bupivacaine USG Supraclavicular Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eslam Ayman Mohamed Shawki (Other)
Responsible Party: Sponsor-Investigator, Eslam Ayman Mohamed Shawki, Lecturer of anesthesia, SICU & Pain Management, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DexSupraClav
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Dexamethasone; Supraclavicular Brachial Plexus Block
Keywords: dexamethasone; supraclavicular brachial plexus block; ultrasound
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to 4 groups:
  * Group A: N-12 will receive a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 0.5ml (2mg) Dexamethasone, 1.5ml Normal saline.
  * Group B: N-12 will receive a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 1ml (4mg) Dexamethasone, 1ml Normal saline.
  * Group C: N-12 will receive a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 2ml (8mg) Dexamethasone.
  * Group Control: N-12 will receive a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 2ml Normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and the attending anesthetist who will manage the patient intra-operatively and perform the block, will be blinded to the patient group allocation All recorded values will be obtained by personnel blinded to the group allocation of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): N-12 Ultrasound guided supraclavicular brachial plexus block will be preformed using a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 0.5ml (2mg) Dexamethasone, 1.5ml Normal saline.
  Interventions: Procedure: Ultrasound guided supraclavicular brachial plexus block; Drug: Dexamethasone
- Group B (Active Comparator): N-12 Ultrasound guided supraclavicular brachial plexus block will be preformed using a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 1ml (4mg) Dexamethasone, 1ml Normal saline.
  Interventions: Procedure: Ultrasound guided supraclavicular brachial plexus block; Drug: Dexamethasone
- Group C (Active Comparator): N-12 Ultrasound guided supraclavicular brachial plexus block will be preformed using a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 2ml (8mg) Dexamethasone.
  Interventions: Procedure: Ultrasound guided supraclavicular brachial plexus block; Drug: Dexamethasone
- Group Control (Active Comparator): N-12 Ultrasound guided supraclavicular brachial plexus block will be preformed using a total volume solution of 20ml: 18ml Bupivacaine 0.5%, 2ml Normal saline.
  Interventions: Procedure: Ultrasound guided supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Ultrasound guided supraclavicular brachial plexus block — ultrasound guided Supraclavicular brachial plexus block
Drug: Dexamethasone — Various doses of Dexamethasone (2, 4 & 8 mg) to be used as an Adjuvant to Local anesthetic drugs
  Other Names: Decadron
  Arms: Group A; Group B; Group C

SUMMARY:
A dose-ranging study to test various doses of Dexamethasone (2, 4 & 8 mg) to be used as an adjuvant to Local anesthetic drugs in ultrasound guided low volume Supraclavicular brachial plexus block to find the best balance between valuable effects (mainly duration of analgesic Effect) and side-effects (mainly increased random blood sugar levels)

DETAILED DESCRIPTION:
Brachial plexus nerve blocks (BPBs) for upper extremity surgery provide superior analgesia and reduce opioid consumption. Supraclavicular block anesthetizes the brachial plexus where it is in its most compact form, thus providing a complete and reliable block for upper extremity surgery. Ultrasound guided single injection (SI) and triple injection (TI) techniques were found to provide the same degree of surgical anesthesia at 30 minutes while the TI technique needed more time to perform.

Many studies were conducted to examine the effect of perineural Dexamethasone as a local anesthetic adjuvant in low volume peripheral nerve blocks were it was found to increase the mean duration of analgesia (sensory block) with short, medium and long acting local anesthetics as well as the duration of motor blockade, with a reduction in pain scores at rest during the intermediate (8-12 h) and late (24 h) postoperative periods and in movement at all times. At 24 postoperative hours, cumulative morphine consumption and the rate of nausea or vomiting were also reduced without any reported related serious adverse effects, also the value of its concomitant intravenous use in prolonging the duration of analgesia after regional blocks was studied with promising results that can sometimes be compared to the perineural route but more short-lived and associated with higher increase in blood glucose levels. Dexamethasone's mechanism of action may result from decreased nociceptive C-fibre activity via a direct effect on glucocorticoid receptors and inhibitory effect on potassium channels.(8) Other authors suggest a local vasoconstrictive effect, resulting in reduced local anaesthetic absorption or a systemic anti-inflammatory effect following vascular uptake of the drug.

A debate exists whether perineural corticosteroids are harmful or not, but reports of neurotoxicity seem to be related mainly to the preservative benzyl alcohol and the vehicle polyethylene glycol found in some preparations, also may be related to the presence of insoluble steroid particulate matter in the injectate. Dexamethasone is non-particulate and can be found in a preservative-free formulation. In addition, no significant long-term electrophysiological, behavioural or histological effects for corticosteroids were identified on rat sciatic nerve tissue even some data suggest dexamethasone may actually be neuroprotective. In reality, perineural corticosteroid injections with and without preservative are widely used throughout the world.

Various doses of Dexamethasone were used in local anaesthetic mixtures in regional blocks in various studies, including 4, 5, 8 and 10 mg. In a recent review & meta-analysis by E. Albrecht and his colleagues, sub-group analysis revealed no association between the total dose of perineural Dexamethasone and the mean increase in duration of analgesia showing that Dose-finding studies are needed to better define the optimal balance between dose, effects and side-effects, particularly at doses lower than 4 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgeries in the upper limb (arm, forearm or hand)

Exclusion Criteria:

* Coagulopathies (with prothrombin concentration less than 60% or INR more than 1.5)
* In-ability to postpone anti-coagulation medications.
* Infection or injury or a lesion at the block site.
* Suspected cervical vertebral column injury necessitating using a neck collar.
* A compromised lung on the contralateral side of the block (Pneumothorax, hemothorax or Pneumonectomy).
* Traumatic vascular injuries or operative interventions (Surgical harvesting) involving arteries of the upper limb on the operative side.
* Patients with communication difficulties.
* Hypersensitivity to local anesthetics and/or Dexamethasone.
* Patients on perioperative intravenous (IV) steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | 24 hours
  The time between injection of Local anesthetic mixture during performing the block and time of administration of the first dose of rescue analgesia at VAS equal or more than 4

SECONDARY OUTCOMES:
Duration of motor block | 24 hours
  The time between injection of Local anesthetic mixture during performing the block and regaining full motor power in the distribution of all 4 nerves represented by score 6 on Modified Lovett rating scale
Patient Satisfaction score | 24 hours
  A point on a 10 point numeric scale where 0 is very dissatisfied and 10 very satisfied one time at the end of the first postoperative 24 hours
Random Blood glucose levels | 24 hours
  Random blood glucose level readings will be obtained from the patient using fast strip test (ACCU-CHEK.) First, upon arrival to the operating theatre, then at the end of the operation then every 8 hours in the first 24 hours postoperatively
Incidence of PONV | 24 hours
  Incidence of postoperative nausea and vomiting
Incidence of complications | 24 hours
  Incidence of Pneumothorax, Nerve injury, Haematoma formation, Intravascular injection

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo University teaching hospitals (Kasr Alainy), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Neal JM, Hebl JR, Gerancher JC, Hogan QH. Brachial plexus anesthesia: essentials of our current understanding. Reg Anesth Pain Med. 2002 Jul-Aug;27(4):402-28. doi: 10.1053/rapm.2002.34377. No abstract available. PMID 12132064
- [Background] Al Harbi M, Kaki AM, Kamal A, El-Dawlatly A, Daghistani M, El Tahan MR. A survey of the practice of regional anesthesia in Saudi Arabia. Saudi J Anaesth. 2013 Oct;7(4):367-70. doi: 10.4103/1658-354X.121041. PMID 24348284
- [Background] Rosenfeld DM, Ivancic MG, Hattrup SJ, Renfree KJ, Watkins AR, Hentz JG, Gorlin AW, Spiro JA, Trentman TL. Perineural versus intravenous dexamethasone as adjuncts to local anaesthetic brachial plexus block for shoulder surgery. Anaesthesia. 2016 Apr;71(4):380-8. doi: 10.1111/anae.13409. Epub 2016 Feb 22. PMID 26899862
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Result] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271